CLINICAL TRIAL: NCT07294391
Title: The Preliminary Efficacy and Safety of Intra-Arterial Albumin as Adjunct to Mechanical Thrombectomy in Acute Ischemic Stroke：Dual-Center, Prospective, Open-Label, Endpoint-Blinded, Randomized Controlled Clinical Trial
Brief Title: The Preliminary Efficacy and Safety of Intra-Arterial Albumin as Adjunct to Mechanical Thrombectomy in Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Huanhu Hospital (Other)
Collaborators: The First Hospital of Qinhuangdao (Other Government)
Responsible Party: Principal Investigator, Ming Wei, PhD, Tianjin Huanhu Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJHH_WM_20251125
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke From Large Vessel Occlusion
Keywords: Acute ischemic stroke; large vessel occlusion; mechanical thrombectomy; albumin; neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: independent Imaging Core Laboratory
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Albumin Group (Experimental): Subjects assigned to the albumin treatment group after achieving successful recanalization (eTICI ≥ 2b) confirmed by DSA post-thrombectomy will receive a 20% human albumin solution at a dose of 0.60 g/kg. The solution will be administered as a constant-rate infusion into the proximal internal carotid artery over 20 minutes. Vital signs and potential infusion-related reactions must be closely monitored throughout the procedure.
  Interventions: Drug: Human serum albumin infusion 20%
- Control Group (No Intervention): Subjects in the control group who have achieved successful recanalization (eTICI ≥ 2b) as confirmed by DSA following mechanical thrombectomy will not receive the investigational infusion and will undergo standard medical management only.

INTERVENTIONS:
Drug: Human serum albumin infusion 20% — 20% human albumin solution at a dose of 0.60 g/kg will be administered as a constant-rate infusion into the proximal internal carotid artery over 20 minutes.
  Arms: Albumin Group

SUMMARY:
Albumin-assisted therapy has demonstrated good safety and potential neuroprotective effects following mechanical thrombectomy. To further systematically evaluate its efficacy and safety, we are conducting a Phase IIa clinical trial of intra-arterial albumin administration combined with mechanical thrombectomy in patients with acute ischemic stroke. This is a double-center, prospective, open-label, endpoint-blinded, randomized controlled trial designed to preliminarily assess the efficacy and safety of intra-arterial infusion of 20% human albumin after successful recanalization in patients with acute ischemic stroke caused by anterior circulation large-vessel occlusion who undergo mechanical thrombectomy. A total of 60 patients will be enrolled and randomized in a 1:1 ratio by dynamic minimization into two groups: the albumin group (0.6 g/kg of 20% human albumin solution plus mechanical thrombectomy) and the control group (mechanical thrombectomy alone).

The primary objective of this study is to preliminarily evaluate whether intra-arterial infusion of 0.6 g/kg of 20% human albumin via the internal carotid artery immediately after achieving successful recanalization (eTICI ≥ 2b) can reduce infarct volume compared with mechanical thrombectomy alone in patients with anterior circulation large-vessel occlusion who undergo standard mechanical thrombectomy. The secondary objective is to assess the safety and feasibility of intra-arterial infusion of 0.6 g/kg of 20% human albumin immediately after successful recanalization in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥ 18 years; 2.ICA or MCA-M1 occlusion, confirmed by preoperative CTA/MRA/DSA. ICA occlusion can be cervical or intracranial, with or without tandem MCA lesions; Treated with EVT resulting in recanalization ((expanded Thrombolysis in Cerebral Infarction [eTICI] 2b-3); 3.Baseline NIHSS scores ≥ 6; 4.Baseline ASPECTS ≥6 on non-contrast CT; 5.The time from stroke onset/last seen well to arterial puncture is within 24 hours; 6.No significant pre-stroke disability (pre-stroke mRS ≤2); 7.Signed informed consent from the patient or the legally authorized representative

Exclusion Criteria:

* 1.Presence of intracranial hemorrhage on head CT or MRI； 2.Midline shift with significant mass effect on head CT or MRI； 3.History of heart failure or severe cardiovascular disease, including but not limited to pulmonary hypertension, pericardial effusion, etc； 4.Arrhythmia accompanied by hemodynamic instability； 5.Symptoms or electrocardiographic evidence of acute myocardial infarction upon admission； 6.Acute or chronic renal failure (serum creatinine >2.0 mg/dL)； 7.Severe anemia (hematocrit <32%)； 8.Known allergy to albumin or blood products； 9.Pregnant women； 10.Persistent blood pressure ≥180/100 mmHg prior to albumin infusion； 11.Concurrent participation in another clinical trial； 12.Life expectancy of less than 3 months； 13.Coexisting severe pulmonary diseases such as Chronic Obstructive Pulmonary Disease, pulmonary fibrosis, pleural effusion, pulmonary hypertension, or acute respiratory distress syndrome； 14.Any other condition that, in the opinion of the investigator, makes the patient unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Growth in infarct volume at 24 (±6) hours after randomization compared to baseline | at 24 (±6) hours after randomization
  MRI-DWI

SECONDARY OUTCOMES:
Proportion of favorable functional outcome at 90 (±14) days, defined as mRS 0-2 | at 90 (±14) day after randomizatio
  mRS
Infarct volume at 24 (±6) hours | at 24 (±6) hours after randomization
  MRI-DWI
Proportion of excellent functional at 90 (±14) days, defined as mRS 0-1 | at 90 (±14) day after randomization
  mRS
mRS score at 90 (±14) days | at 90 (±14) days after randomization
  mRS
Vessel recanalization at 24 (±6) hours | at 24 (±6) hours after randomization
  CTA or MRA or DSA
NIHSS score at 24 (±6) hours | at 24 (±6) hours after randomization
  NIHSS
NIHSS score at 7 (±1) days/at discharge | at 7 (±1) days/at discharge after randomization
  NIHSS
EQ-5D-5L at 90 (±14) days | at 90 (±14) days after randomization
  EQ-5D-5L
Proportion of Barthel Index ≥95 at 90 (±14) days | at 90 (±14) days after randomization
  Barthel Index
Incidence of all-cause death within 90 (±14) days | at 90 (±14) days after randomization
  all-cause death
Incidence of symptomatic intracranial hemorrhage within 24 (±6) hours | at 24 (±6) hours after randomization
  according to the modified Heidelberg Bleeding Classification
Incidence of intracranial hemorrhage within 24 (±6) hours | at 24 (±6) hours after randomization
  all-cause
Incidence of serious adverse events within 90 (±14) days | at 90 (±14) days after randomization
  serious adverse events
Incidence of adverse events within 90 (±14) days | at 90 (±14) days after randomization
  adverse events
Proportion of early neurological deterioration at 24 hours | at 24 hours after randomization
  defined as ≥ 4-point increase in NIHSS score from baseline
Proportion of severe disability at 90 (±14) days | at 90 (±14) days after randomization
  defined as mRS 4-6
Incidence of albumin infusion-associated adverse event within 24 (± 6) hours | at 24 (± 6) hours after randomization
  albumin infusion-associated adverse event

OTHER OUTCOMES:
Blood levels of albumin and BNP at 24 (±6) hours after randomization | at 24 (±6) hours after randomization
  albumin and BNP
Blood levels of albumin and BNP at 7 (±1) days after randomization or at discharge (whichever occurs first) | at 7 (±1) days after randomization or at discharge (whichever occurs first)
  albumin and BNP
The along the perivascular space (ALPS) index at 24 (±6) hours after randomization | at 24 (±6) hours after randomization
  along the perivascular space index

IPD SHARING:
Plan to Share IPD: Undecided